CLINICAL TRIAL: NCT06982755
Title: Effect of Acupuncture on Early Analgesia of Non-traumatic Acute Abdomen is Discussed Based on the Experience of Sanli Acupoint for Du-fu Diseases :A Prospective Randomized Controlled pRCT Study
Brief Title: Acupuncture Versus Compound Diclofenac Sodium for Pain Relief in Non-Traumatic Acute Abdominal
Acronym: ACU-NTAA
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Hunan University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A2024021
Record Dates: First submitted 2025-04-24; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Acute Abdominal Pain; Acupuncture Therapy; Acupuncture; Opioids
Keywords: Acute abdominal pain; Non-Traumatic Acute Abdomen; Non-traumatic acute abdomen early analgesia; Acupuncture therapy; Acupuncture; Zusanli point, ST36; Diclofenac sodium; Emergency environment; Opioids; Non-steroidal anti-inflammatory drugs ，NSAIDs; Acetaminophen
MeSH Terms: conditions — Abdomen, Acute | interventions — Acupuncture Therapy

STUDY DESIGN:
Masking Description: This study is classified as exploratory research. This designation is due to the specialized techniques required for acupuncture and sham acupuncture, as well as the significant differences in intervention methods between acupuncture and intramuscular injection of diclofenac sodium. Given these factors, a double-blind approach was not feasible in this study. To minimize open-label bias, the principal investigators, operators, outcome assessors, data collectors, and statistical analysts will act independently in all aspects of the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- acupuncture group (Active Comparator): acupuncture at Zusanli (ST36)
  Interventions: Procedure: acupuncture; Drug: compound diclofenac sodium; Combination Product: acupuncture combined with compound diclofenac sodium; Combination Product: placebo
- compound diclofenac sodium group (Active Comparator): intramuscular injection of compound diclofenac sodium injection
  Interventions: Procedure: acupuncture; Drug: compound diclofenac sodium; Combination Product: acupuncture combined with compound diclofenac sodium; Combination Product: placebo
- acupuncture combined with compound diclofenac sodium group (Experimental): acupuncture at Zusanli (ST36) and intramuscular injection of compound diclofenac sodium injection
  Interventions: Procedure: acupuncture; Drug: compound diclofenac sodium; Combination Product: acupuncture combined with compound diclofenac sodium; Combination Product: placebo
- placebo group (Placebo Comparator): superficial acupuncture at Zusanli (ST36) and intramuscular injection of normal saline
  Interventions: Procedure: acupuncture; Drug: compound diclofenac sodium; Combination Product: acupuncture combined with compound diclofenac sodium; Combination Product: placebo

INTERVENTIONS:
Procedure: acupuncture — acupuncture at Zusanli (ST36); sample size: 44
Drug: compound diclofenac sodium — intramuscular injection of compound diclofenac sodium injection; sample size: 44
  Other Names: compound Diclofenac Sodium Injection
Combination Product: acupuncture combined with compound diclofenac sodium — acupuncture at Zusanli (ST36) and intramuscular injection of compound diclofenac sodium injection; sample size: 44
Combination Product: placebo — superficial acupuncture at Zusanli (ST36) and intramuscular injection of normal saline; sample size: 44

SUMMARY:
The investigators designed this clinical study to evaluate the efficacy and safety of semi-standardized acupuncture and moxibustion combined with compound diclofenac sodium injection in the emergency department (ED) compared with acupuncture or compound diclofenac sodium injection alone.

DETAILED DESCRIPTION:
This study is a prospective, parallel-controlled, open-label randomized controlled trial (RCT). The Numeric Rating Scale (NRS) was used to assess pain intensity. The primary outcome measure was the difference in pain response rates between the combined intervention group, the acupuncture-only group, and the diclofenac sodium combination group at 10 minutes post-treatment compared to baseline. Secondary outcomes included treatment response rates, NRS scores, pain recurrence rates, rescue medication rates, and adverse events at each observation time point across the three groups. Additionally, a placebo group was included to exploratorily assess the placebo effect of the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. The diagnostic criteria of NTAA were as follows: ① abdominal pain was the main symptom; ② The onset time was less than 1 week; ③ The cause of abdominal pain could be traced to intra-abdominal abdominal wall chest or systemic diseases;
2. Patients with NRS scores ≥4 (mild pain and above) were evaluated before inclusion; （3）16 years < age <75 years;

（4）Those who were considered not to need surgery within 2 hours after initial assessment by a specialist.

Exclusion Criteria:

Participants meeting any of the following criteria were excluded from the study:

1. Acute abdomen caused by trauma;
2. Super sudden diseases (e.g. acute myocardial infarction rupture of abdominal aortic aneurysm pulmonary embolism aortic dissection pericardial tamponade);
3. Emergent conditions requiring surgical treatment within 3 hours (e.g. rupture of liver cancer ectopic pregnancy ischemic bowel disease severe acute cholangitis peritonitis with septic shock);
4. Extremely severe pain (NRS ≥ 8) with an undetermined diagnosis and requiring further assessment for a super sudden disease;
5. Inability to select acupuncture points due to skin injury or ulceration at Zusanli (ST36) on the lower limb;
6. Induration or infection at the hip injection site;
7. Patients with altered consciousness mental illness other severe chronic diseases or those who are unlikely to cooperate with acupuncture treatment;
8. Contraindications to Western medicine:

   * Known allergies to diclofenac sodium or acetaminophen; ②History of asthma urticaria or allergic reactions induced by aspirin or other NSAIDs.

     * Undergoing coronary artery bypass grafting (CABG) surgery. ④History of gastrointestinal bleeding or perforation following non-steroidal anti-inflammatory drugs (NSAIDs).

       * Active gastrointestinal ulcers or bleeding or a history of recurrent ulcers or bleeding.

         * Severe heart failure.
9. Use of any pain medication or acupuncture within the past 6 hours;
10. Previous participation in this study;
11. Pregnant or lactating individuals.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain response rate | at 10 minutes after analgesia
  Using the Numeric Rating Scale (NRS) score evaluate the proportion of individuals within the group who achieved a therapeutic index of ≥50% at the 10th minute post-treatment compared to baseline

SECONDARY OUTCOMES:
The utilization rate of rescue drugs | within 1 hour to 1 day post-analgesia
  If the subject still experiences intolerable pain (NRS ≥ 4) after 1 hour of treatment or following supplemental treatment, additional analgesic medications such as Rotundine or Dezocine shall be administered. Furthermore, subjects who still exhibit "severe pain" after 1 hour of treatment will be given rescue analgesic medication: Pethidine Hydrochloride Injection, 25 mg, intramuscularly (to be prescribed by a supervising physician with the qualifications to prescribe narcotic drugs).
Expectations with the intervention | baseline
  In this study, a Likert scale was utilized to construct a specialized questionnaire aimed at assessing patients' expectations of the intervention. The questionnaire consists of four items designed to evaluate patients' anticipations regarding the intervention's efficacy in alleviating symptoms, its onset of action, potential side effects, and its impact on quality of life. Each item is scored on a five-point scale, ranging from 1 (strongly disagree) to 5 (strongly agree). At baseline, the ratings for each item were determined according to the personal expectations of the patients. To provide a comprehensive reflection of patients' overall expectations of the intervention, each item is assigned equal weight in the total score calculation. The scores of the four items are summed to yield a total score, which quantifies patients' overall expectations of the intervention.
Satisfaction with the intervention | at 1 day after analgesia
  In this study, a Likert scale was employed to develop a specialized questionnaire designed to assess patient satisfaction with the intervention. The questionnaire comprehensively evaluates patient satisfaction across multiple dimensions, including satisfaction with the treatment process, experience of side effects, and overall satisfaction. Each dimension is rated on a five-point scale, ranging from 1 (strongly disagree) to 5 (strongly agree). The items in the questionnaire were rated by patients based on their actual experiences on the first day after the intervention. To provide a comprehensive reflection of patients' overall satisfaction with the intervention, each item carries equal weight in the total score calculation. The scores of all items are summed to yield a total score, which quantifies the patients' overall satisfaction with the intervention.
Numeric Rating Scale (NRS) score | at 0, 1, 5, 10, 20, 30, and 60 minutes, and at 1 and 3 days post-analgesia
  Numeric Rating Scale
Recurrence rate of pain | at 1 day after analgesia
  Recurrence rate of pain within 1 day in the four groups: NRS score ≤2 after the initial intervention pain recurrence within 1 day and occurrence of NRS score ≥4.

OTHER OUTCOMES:
Avatar Incidence of adverse events | through study completion, an average of 3 days
  During the entire treatment period and follow-up period: Adverse events were evaluated immediately after the intervention, at 0, 1, 5, 10, 20, 30, and 60 minutes after the treatment, and during the follow-up periods on the first and third days after the intervention. The frequency of adverse events in each group was recorded, and the proportion of adverse events was calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Zhong Feng, Ph.D., Study Director — Hunan University of Traditional Chinese Medicine